CLINICAL TRIAL: NCT01966770
Title: Clinical Evaluation of Hydrogels vs Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-44
Record Dates: First submitted 2013-10-15; First posted 2013-10-22 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Pair 1 (ocufilcon D / ocufilcon D) (Active Comparator): Randomized to contra lateral lens pair 1 (ocufilcon D hydrogel / ocufilcon D hydrogel)
  Interventions: Device: Pair 1 (ocufilcon D / ocufilcon D)
- Pair 2 (ocufilcon D / enfilcon A) (Active Comparator): Randomized to contra lateral lens pair 2 (ocufilcon D hydrogel / enfilcon A silicone)
  Interventions: Device: Pair 2 (ocufilcon D / enfilcon A)
- Pair 3 (ocufilcon D / comfilcon A) (Active Comparator): Randomized to contra lateral lens pair 3 (ocufilcon D hydrogel / comfilcon A silicone)
  Interventions: Device: Pair 3 (ocufilcon D / comfilcon A)
- Pair 4 (methafilcon A / methafilcon A) (Active Comparator): Randomized to contra lateral lens pair 4 (methafilcon A hydrogel sphere / methafilcon A hydrogel asphere)
  Interventions: Device: Pair 4 (methafilcon A / methafilcon A)
- Pair 5 (methafilcon A / comfilcon A) (Active Comparator): Randomized to contra lateral lens pair 5 (methafilcon A hydrogel / comfilcon A silicone)
  Interventions: Device: Pair 5 (methafilcon A / comfilcon A)
- Pair 6 (omafilcon A / comfilcon A) (Active Comparator): Randomized to contra lateral lens pair 6 (omafilcon A hydrogel / comfilcon A silicone)
  Interventions: Device: Pair 6 (omafilcon A / comfilcon A)

INTERVENTIONS:
Device: Pair 1 (ocufilcon D / ocufilcon D) — Randomized to contra lateral lens pair 1 (ocufilcon D hydrogel / ocufilcon D hydrogel)
  Arms: Pair 1 (ocufilcon D / ocufilcon D)
Device: Pair 2 (ocufilcon D / enfilcon A) — Randomized to contra lateral lens pair 2 (ocufilcon D hydrogel / enfilcon A silicone)
  Arms: Pair 2 (ocufilcon D / enfilcon A)
Device: Pair 3 (ocufilcon D / comfilcon A) — Randomized to contra lateral lens pair 3 (ocufilcon D hydrogel / comfilcon A silicone)
  Arms: Pair 3 (ocufilcon D / comfilcon A)
Device: Pair 4 (methafilcon A / methafilcon A) — Randomized to contra lateral lens pair 4 (methafilcon A hydrogel sphere / methafilcon A hydrogel asphere)
  Arms: Pair 4 (methafilcon A / methafilcon A)
Device: Pair 5 (methafilcon A / comfilcon A) — Randomized to contra lateral lens pair 5 (methafilcon A hydrogel / comfilcon A silicone)
  Arms: Pair 5 (methafilcon A / comfilcon A)
Device: Pair 6 (omafilcon A / comfilcon A) — Randomized to contra lateral lens pair 6 (omafilcon A hydrogel / comfilcon A silicone)
  Arms: Pair 6 (omafilcon A / comfilcon A)

SUMMARY:
The aim of this fitting study is to evaluate the clinical performance of different hydrogel and silicone hydrogel contact lenses.

DETAILED DESCRIPTION:
This is a 20-subject, double masked, randomized, contra lateral, 2-day non-dispensing fitting trial.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft contact lens wearer
* Has a cl spherical prescription between -1.00 and -6.00 (inclusive)
* Has a spectacle cylinder up to 0.75D (diopter) in each eye
* Is correctable to a visual acuity of 20/25 or better in both eyes
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter
* Is willing to comply with the wear schedule
* Is willing to comply with the visit schedule

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has never worn contact lenses before
* Currently wears rigid gas permeable contact lenses
* Has a history of not achieving comfortable contact lens wear (5 days per week; > 8 hours/day)
* Has a contact lens prescription outside the range of -1.00 to -6.00D
* Has a spectacle cylinder ≥ 1.00D of cylinder in either eye
* Has best corrected spectacle distance vision worse than 20/25 in either eye
* Has any systemic or topical medications that will affect ocular health
* Has any ocular pathology or severe insufficiency of lacrimal secretion
* Has persistent, clinically significant corneal or conjunctival staining
* Has active neovascularization or any central corneal scars
* Is aphakic
* Is presbyopic
* Has undergone corneal refractive surgery
* Is participating in any other type of eye related conical or research study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng Lin, OD PhD FAAO, Principal Investigator — CRC-UC Berkeley
Locations (1):
- University of California, Berkeley Clinical Research Center (UCB-CRC), Berkeley, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study Group: All participants were habitual contact lens wearers and all participants wore Day 1 followed by Day 2 lenses
Period: Overall Study
Arm/Group | Overall Study Group
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All particpants wore Day 1 followed by Day 2 lenses
Arm/Group | Overall Study Group
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 10
  Non-Asian | 10
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (VA) logMAR (Habitual Lenses)
Description: Assessment of high contrast distance visual acuity (VA). Collected at baseline with subject wearing habitual lens prior to dispense of study lens. (logMAR)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: LogMar
Groups:
- Habitual Lens: Subjects presented wearing habitual lenses prior to dispense of study lenses.
Arm/Group | Habitual Lens
Number analyzed (Participants) | 20
LogMar | -0.06 (0.08)

2. Primary Outcome: Visual Acuity (VA) logMAR (Study Lenses)
Description: Assessment of high contrast distance visual acuity (VA). Collected at dispense of study lens. (logMAR)
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- B55 PREMIER ASPHERE LENS: Subjects wore contralateral lenses. Biomedics 55 Asphere (B55 PREMIER ASPHERE LENS) in one eye and Biomedics 55 Sphere (B55 SPHERE LENS) in the other.
- B55 SPHERE LENS: Subjects wore contralateral lenses. Biomedics 55 Sphere (B55 SPHERE LENS) in one eye and either Biomedics 55 Asphere (B55 PREMIER ASPHERE LENS) or Biofinity (BF SPHERE LENS) or Avaira (AV SPHERE LENS) in the other.
- BF SPHERE LENS: Subjects wore contralateral lenses. Biofinity (BF SPHERE LENS) in one eye and Biomedics 55 Sphere (B55 SPHERE LENS) in the other.
- AV SPHERE LENS: Subjects wore contralateral lenses. Avaira (AV SPHERE LENS) in one eye and Biomedics 55 Sphere (B55 SPHERE LENS) in the other.
- PCM SPHERE LENS: Subjects wore contralateral lenses. Proclear Monthly (PCM SPHERE LENS) in one eye and Biofinity (BF SPHERE LENS) in the other. Collected at study lens dispense.
- F55 SPHERE LENS: Subjects wore contralateral lenses. Frequency 55 Sphere (F55 SPHERE LENS) in one eye and either Frequency 55 Asphere (F55 ASPHERE LENS) or Biofinity (BF SPHERE LENS) in the other.
- F55 ASPHERE LENS: Subjects wore contralateral lenses. Frequency 55 Asphere (F55 ASPHERE LENS) in one eye and Frequency 55 Sphere (F55 SPHERE LENS) in the other.
Arm/Group | B55 PREMIER ASPHERE LENS | B55 SPHERE LENS | BF SPHERE LENS | AV SPHERE LENS | PCM SPHERE LENS | F55 SPHERE LENS | F55 ASPHERE LENS
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20
LogMAR | -0.13 (0.06) | -0.11 (0.07) | -0.13 (0.06) | -0.12 (0.06) | -0.13 (0.07) | -0.11 (0.08) | -0.13 (0.07)

3. Primary Outcome: Comfort Contact Lens Insertion (Day 1 Study Lenses)
Description: Participant rating of comfort upon contact lens insertion. Collected after insertion at Day 1 for each lens . (0-100, 0=cannot be worn causes pain, 100=cannot be felt ever)
Time Frame: Day 1 - Insertion
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- B55 SPHERE LENS P1; B55 PREMIER ASPHERE LENS P1: Subjects wore contralateral lenses. Biomedics 55 Sphere (B55 SPHERE LENS) in one eye and Biomedics 55 Asphere (B55 PREMIER ASPHERE LENS) in the other.
- B55 SPHERE LENS P2; AV SPHERE LENS P2: Subjects wore contralateral lenses. Biomedics 55 Sphere (B55 SPHERE LENS) in one eye and Avaira (AV SPHERE LENS) in the other.
- B55 SPHERE LENS P3; BF SPHERE LENS P3: Subjects wore contralateral lenses. Biomedics 55 Sphere (B55 SPHERE LENS) in one eye and Biofinity (BF SPHERE LENS) in the other.
Arm/Group | B55 SPHERE LENS P1 | B55 PREMIER ASPHERE LENS P1 | B55 SPHERE LENS P2 | AV SPHERE LENS P2 | B55 SPHERE LENS P3 | BF SPHERE LENS P3
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
units on a scale | 92 (8) | 95 (6) | 95 (7) | 97 (5) | 95 (8) | 96 (6)

4. Primary Outcome: Comfort Contact Lens 30 Minutes Wear (Day 1 Study Lenses)
Description: Participant rating of comfort after contact lens settling. Collected at 30 minutes wear for each lens. (0-100, 0=cannot be worn causes pain, 100=cannot be felt ever)
Time Frame: Day 1 - 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | B55 SPHERE LENS P1 | B55 PREMIER ASPHERE LENS P1 | B55 SPHERE LENS P2 | AV SPHERE LENS P2 | B55 SPHERE LENS P3 | BF SPHERE LENS P3
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
units on a scale | 97 (1.8) | 96 (1.3) | 96 (1.6) | 96 (1.1) | 96 (1.8) | 95 (1.3)

5. Primary Outcome: Comfort Contact Lens Insertion (Day 2 Study Lenses)
Description: Participant rating of comfort upon contact lens insertion. Collected after insertion at Day 2 for each lens . (0-100, 0=cannot be worn causes pain, 100=cannot be felt ever
Time Frame: Day 2 - Insertion
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- F55 SPHERE LENS P1; F55 ASPHERE LENS P1: Subjects wore contralateral lenses. Frequency 55 Sphere (F55 SPHERE LENS) in one eye and Frequency 55 Asphere (F55 ASPHERE LENS) in the other.
- F55 SPHERE LENS P2; BF SPHERE LENS P2: Subjects wore contralateral lenses. Frequency 55 Sphere (F55 SPHERE LENS) in one eye and Biofinity (BF SPHERE LENS) in the other.
- PCM SPHERE LENS P3; BF SPHERE LENS P3: Subjects wore contralateral lenses. Proclear Monthly (PCM SPHERE LENS) in one eye and Biofinity (BF SPHERE LENS) in the other.
Arm/Group | F55 SPHERE LENS P1 | F55 ASPHERE LENS P1 | F55 SPHERE LENS P2 | BF SPHERE LENS P2 | PCM SPHERE LENS P3 | BF SPHERE LENS P3
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
units on a scale | 94 (14) | 92 (16) | 93 (14) | 96 (8.0) | 94 (10) | 97 (9.0)

6. Primary Outcome: Comfort Contact Lens 30 Minutes Wear (Day 2 Study Lenses)
Description: Participant rating of comfort upon contact lens insertion. Collected after 30 minutes of wear at Day 2 for each lens . (0-100, 0=cannot be be worn causes pain, 100=cannot be felt ever
Time Frame: Day 2 - 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | F55 SPHERE LENS P1 | F55 ASPHERE LENS P1 | F55 SPHERE LENS P2 | BF SPHERE LENS P2 | PCM SPHERE LENS P3 | BF SPHERE LENS P3
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
units on a scale | 96 (6.0) | 93 (13) | 94 (10) | 96 (6.0) | 97 (7.0) | 98 (3.0)

7. Primary Outcome: Comfort Preference Contact Lens Insertion (Day 1 Study Lenses - Pair 1)
Description: Participant rating of comfort preference upon contact lens insertion of pair 1. Collected at insertion for each lens. Percent of participants that strongly prefer lens or have No Preference. (forced choice preference for right or left eye; Strongly Prefer Left, Slightly Prefer Left, No Preference, Slightly Prefer Right, Strongly Prefer Right)
Time Frame: Day 1 - Insertion
Measure: Number; unit: percentage of participants
Groups:
- B55 SPHERE LENS P1 / B55 PREMIER ASPHERE LENS P1: Subjects wore contralateral lenses. Pair 1 Biomedics 55 Sphere (B55 SPHERE LENS) in one eye and Biomedics 55 Asphere (B55 PREMIER ASPHERE LENS) in the other.
Arm/Group | B55 SPHERE LENS P1 / B55 PREMIER ASPHERE LENS P1
Number analyzed (Participants) | 20
percentage of participants
  B55 SPHERE LENS P1 | 5
  B55 PREMIER ASPHERE LENS P1 | 35
  No Preference | 60

8. Primary Outcome: Comfort Preference Contact Lens Insertion (Day 1 Study Lenses - Pair 2)
Description: Participant rating of comfort preference upon contact lens insertion of pair 2. Collected at insertion for each lens. Percent of participants that strongly prefer lens or have No Preference. (forced choice preference for right or left eye; Strongly Prefer Left, Slightly Prefer Left, No Preference, Slightly Prefer Right, Strongly Prefer Right)
Time Frame: Day 1 Insertion
Measure: Number; unit: percentage of participants
Groups:
- B55 SPHERE LENS P2 / AV SPHERE LENS P2: Subjects wore contralateral lenses. Pair 2 Biomedics 55 Sphere (B55 SPHERE LENS P2) in one eye and Avairia sphere (AV SPHERE LENS P2) in the other.
Arm/Group | B55 SPHERE LENS P2 / AV SPHERE LENS P2
Number analyzed (Participants) | 20
percentage of participants
  B55 SPHERE LENS P2 | 0
  AV SPHERE LENS P2 | 15
  No Preference | 85

9. Primary Outcome: Comfort Preference Contact Lens Insertion (Day 1 Study Lenses - Pair 3)
Description: Participant rating of comfort preference upon contact lens insertion of pair 3. Collected at insertion for each lens. Percent of participants that strongly prefer lens or have No Preference. (forced choice preference for right or left eye; Strongly Prefer Left, Slightly Prefer Left, No Preference, Slightly Prefer Right, Strongly Prefer Right)
Time Frame: Day 1 - Insertion
Measure: Number; unit: percentage of participants
Groups:
- B55 SPHERE LENS P3 / BF SPHERE LENS P3: Subjects wore contralateral lenses. Pair 3 Biomedics 55 Sphere (B55 SPHERE LENS P3) in one eye and Biofinity (BF SPHERE LENS P3) in the other.
Arm/Group | B55 SPHERE LENS P3 / BF SPHERE LENS P3
Number analyzed (Participants) | 20
percentage of participants
  B55 SPHERE LENS P3 | 10
  BF SPHERE LENS P3 | 20
  No Preference | 70

10. Primary Outcome: Comfort Preference Contact Lens 30 Minutes Wear (Day 1 Study Lenses - Pair 1)
Description: Participant rating of comfort preference upon contact lens settling of pair 1. Collected at 30 minutes post settling for each lens. Percent of participants that strongly prefer lens or have No Preference. (forced choice preference for right or left eye; Strongly Prefer Left, Slightly Prefer Left, No Preference, Slightly Prefer Right, Strongly Prefer Right)
Time Frame: Day 1 - 30 minutes
Measure: Number; unit: percentage of participants
Arm/Group | B55 SPHERE LENS P1 / B55 PREMIER ASPHERE LENS P1
Number analyzed (Participants) | 20
percentage of participants
  B55 SPHERE LENS P1 | 10
  B55 PREMIER ASPHERE LENS P1 | 5
  No Preference | 85

11. Primary Outcome: Comfort Preference Contact Lens 30 Minutes Wear (Day 1 Study Lenses - Pair 2)
Description: Participant rating of comfort preference upon contact lens settling of pair 2. Collected at 30 minutes post settling for each lens. Percent of participants that strongly prefer lens or have No Preference. (forced choice preference for right or left eye; Strongly Prefer Left, Slightly Prefer Left, No Preference, Slightly Prefer Right, Strongly Prefer Right)
Time Frame: Day 1 - 30 minutes
Measure: Number; unit: percentage of participants
Arm/Group | B55 SPHERE LENS P2 / AV SPHERE LENS P2
Number analyzed (Participants) | 20
percentage of participants
  B55 SPHERE LENS P2 | 0
  AV SPHERE LENS P2 | 10
  No Preference | 90

12. Primary Outcome: Comfort Preference Contact Lens 30 Minutes Wear (Day 1 Study Lenses - Pair 3)
Description: Participant rating of comfort preference upon contact lens settling of pair 3. Collected at 30 minutes post settling for each lens. Percent of participants that strongly prefer lens or have No Preference. (forced choice preference for right or left eye; Strongly Prefer Left, Slightly Prefer Left, No Preference, Slightly Prefer Right, Strongly Prefer Right)
Time Frame: Day 1 - 30 minutes
Measure: Number; unit: percentage of participants
Arm/Group | B55 SPHERE LENS P3 / BF SPHERE LENS P3
Number analyzed (Participants) | 20
percentage of participants
  B55 SPHERE LENS P3 | 10
  BF SPHERE LENS P3 | 5
  No Preference | 85

13. Primary Outcome: Comfort Preference Contact Lens Insertion (Day 2 Study Lenses - Pair 1)
Description: as for outcome 7
Time Frame: Day 2 - Insertion
Measure: Number; unit: percentage of participants
Groups:
- F55 SPHERE LENS P1 / F55 PREMIER ASPHERE LENS P1: Subjects wore contralateral lenses. Frequency 55 Sphere (F55 SPHERE LENS) in one eye and Frequency 55 Asphere (F55 ASPHERE LENS) in the other.
Arm/Group | F55 SPHERE LENS P1 / F55 PREMIER ASPHERE LENS P1
Number analyzed (Participants) | 20
percentage of participants
  F55 SPHERE LENS P1 | 20
  F55 PREMIER ASPHERE LENS P1 | 10
  No Preference | 70

14. Primary Outcome: Comfort Preference Contact Lens Insertion (Day 2 Study Lenses - Pair 2)
Description: as for outcome 8
Time Frame: Day 2 - Insertion
Measure: Number; unit: percentage of participants
Groups:
- F55 SPHERE LENS P2 / BIOFINITY LENS P2: Subjects wore contralateral lenses. Frequency 55 Sphere (F55 SPHERE LENS) in one eye and Biofinity (BF SPHERE LENS) in the other.
Arm/Group | F55 SPHERE LENS P2 / BIOFINITY LENS P2
Number analyzed (Participants) | 20
percentage of participants
  F55 SPHERE LENS P2 | 10
  BIOFINITY LENS P2 | 15
  No Preference | 75

15. Primary Outcome: Comfort Preference Contact Lens Insertion (Day 2 Study Lenses - Pair 3)
Description: as for outcome 9
Time Frame: Day 2 - Insertion
Measure: Number; unit: percentage of participants
Groups:
- PCM SPHERE LENS P3 / BF SPHERE LENS P3: Subjects wore contralateral lenses. Proclear Monthly (PCM SPHERE LENS) in one eye and Biofinity (BF SPHERE LENS) in the other.
Arm/Group | PCM SPHERE LENS P3 / BF SPHERE LENS P3
Number analyzed (Participants) | 20
percentage of participants
  PCM SPHERE LENS P3 | 5
  BF SPHERE LENS P3 | 15
  No Preference | 80

16. Primary Outcome: Comfort Preference Contact Lens 30 Minutes Wear (Day 2 Study Lenses - Pair 1)
Description: as for outcome 10
Time Frame: Day 2 - 30 minutes
Measure: Number; unit: percentage of participants
Arm/Group | F55 SPHERE LENS P1 / F55 PREMIER ASPHERE LENS P1
Number analyzed (Participants) | 20
percentage of participants
  F55 SPHERE LENS P1 | 10
  F55 PREMIER ASPHERE LENS P1 | 15
  No Preference | 75

17. Primary Outcome: Comfort Preference Contact Lens 30 Minutes Wear (Day 2 Study Lenses - Pair 2)
Description: as for outcome 11
Time Frame: Day 2 - 30 minutes
Measure: Number; unit: percentage of participants
Arm/Group | F55 SPHERE LENS P2 / BIOFINITY LENS P2
Number analyzed (Participants) | 20
percentage of participants
  F55 SPHERE LENS P2 | 10
  BIOFINITY LENS P2 | 10
  No Preference | 80

18. Primary Outcome: Comfort Preference Contact Lens 30 Minutes Wear (Day 2 Study Lenses - Pair 3)
Description: as for outcome 12
Time Frame: Day 2 - 30 minutes
Measure: Number; unit: percentage of participants
Arm/Group | PCM SPHERE LENS P3 / BF SPHERE LENS P3
Number analyzed (Participants) | 20
percentage of participants
  PCM SPHERE LENS P3 | 0
  BF SPHERE LENS P3 | 20
  No Preference | 80

19. Primary Outcome: Lens Fitting Characteristics, Centration (Habitual Lens)
Description: Assessment of habitual lens fitting characteristics for the percentage of lenses with optimal centration. Collected at baseline with subject wearing habitual lens prior to dispense of study lens. (Optimal Centration for Right and Left eyes; Optimum, Decentration Acceptable, Decentration unacceptable)
Time Frame: Baseline
Measure: Number; unit: percentage of eyes
Units Other Than Participants: lens
Arm/Group | Habitual Lens
Number analyzed (Participants) | 20
Number analyzed (lens) | 40
percentage of eyes | 75

20. Primary Outcome: Lens Fitting Characteristics, Tightness (Habitual Lens)
Description: Assessment of habitual lens fitting characteristics. Collected at baseline with subject wearing habitual lens prior to dispense of study lens. Digital push up test. (Continuous scale 0-100%, 0%=falls from cornea without lid support, 50%=optimum, 100%=no movement)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: eyes
Arm/Group | Habitual Lens
Number analyzed (Participants) | 20
Number analyzed (eyes) | 40
percentage | 46 (11)

21. Primary Outcome: Lens Fitting Characteristics, Upgaze Lag and Post-blink Movement (Habitual Lens)
Description: Assessment of habitual lens fitting characteristics. Collected at baseline with subject wearing habitual lens prior to dispense of study lens.(Upgaze Lag and Post-blink Movement in mm)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: lens
Arm/Group | Habitual Lens
Number analyzed (Participants) | 20
Number analyzed (lens) | 40
millimeters
  Upgaze Lag | 0.21 (0.51)
  Post-blink Movement | 0.19 (0.12)

22. Primary Outcome: Lens Fitting Characteristics, Centration (Day 1 Study Lenses)
Description: Assessment of lens fitting characteristics for the percentage of lenses with optimal centration. Collected at 30 minutes after lens settling of study lens. (Optimal Centration for Right and Left eyes; Optimum, Decentration Acceptable, Decentration unacceptable)
Time Frame: Day 1 - 30 minutes
Measure: Number; unit: percentage of lenses
Units Other Than Participants: lens
Arm/Group | B55 SPHERE LENS P1 | B55 PREMIER ASPHERE LENS P1 | B55 SPHERE LENS P2 | AV SPHERE LENS P2 | B55 SPHERE LENS P3 | BF SPHERE LENS P3
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Number analyzed (lens) | 20 | 20 | 20 | 20 | 20 | 20
percentage of lenses | 100 | 100 | 100 | 100 | 100 | 90

23. Primary Outcome: Lens Fitting Characteristics, Push-up Tightness (Day 1 Study Lenses)
Description: Assessment of lens fitting characteristics. Collected at 30 minutes after lens settling of study lens. Digital push up test. (Continuous scale 0-100%, 0%=falls from cornea without lid support, 50%=optimum, 100%=no movement)
Time Frame: Day 1 - 30 minutes
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: lens
Arm/Group | B55 SPHERE LENS P1 | B55 PREMIER ASPHERE LENS P1 | B55 SPHERE LENS P2 | AV SPHERE LENS P2 | B55 SPHERE LENS P3 | BF SPHERE LENS P3
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Number analyzed (lens) | 20 | 20 | 20 | 20 | 20 | 20
percentage | 50 (13) | 48 (13) | 51 (13) | 45 (11) | 52 (16) | 54 (11)

24. Primary Outcome: Lens Fitting Characteristics, Upper Gaze Lag and Post-blink Movement (Day 1 - Study Lenses)
Description: Assessment of lens fitting characteristics. Collected at 30 minutes after lens settling of study lens. (Upgaze Lag and Post-blink Movement in mm)
Time Frame: Day 1 - 30 minutes
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: lens
Arm/Group | B55 SPHERE LENS P1 | B55 PREMIER ASPHERE LENS P1 | B55 SPHERE LENS P2 | AV SPHERE LENS P2 | B55 SPHERE LENS P3 | BF SPHERE LENS P3
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Number analyzed (lens) | 40 | 40 | 40 | 40 | 40 | 40
millimeter
  Upper Gaze Lag | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.05 (0.22) | 0.00 (0.00) | 0.00 (0.00)
  Post-blink Movement | 0.39 (0.43) | 0.39 (0.40) | 0.28 (0.29) | 0.41 (0.28) | 0.27 (0.27) | 0.30 (0.25)

25. Primary Outcome: Lens Fitting Characteristics, Centration (Day 2 Study Lenses)
Description: as for outcome 22
Time Frame: Day 2 - 30 minutes
Measure: Number; unit: percentage of lenses
Units Other Than Participants: lens
Arm/Group | F55 SPHERE LENS P1 | F55 ASPHERE LENS P1 | F55 SPHERE LENS P2 | BF SPHERE LENS P2 | PCM SPHERE LENS P3 | BF SPHERE LENS P3
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Number analyzed (lens) | 20 | 20 | 20 | 20 | 20 | 20
percentage of lenses | 95 | 95 | 95 | 100 | 100 | 100

26. Primary Outcome: Lens Fitting Characteristics, Push-up Tightness (Day 2 Study Lenses)
Description: as for outcome 23
Time Frame: Day 2 - 30 minutes
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: lens
Arm/Group | F55 SPHERE LENS P1 | F55 ASPHERE LENS P1 | F55 SPHERE LENS P2 | BF SPHERE LENS P2 | PCM SPHERE LENS P3 | BF SPHERE LENS P3
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Number analyzed (lens) | 20 | 20 | 20 | 20 | 20 | 20
percentage | 53 (13.4) | 50 (14.9) | 51 (13.5) | 53 (12.3) | 53 (15.2) | 55 (11.7)

27. Primary Outcome: Lens Fitting Characteristics, Upper Gaze Lag and Post-blink Movement (Day 2 Study Lenses)
Description: Assessment of lens fitting characteristics. Collected at 30 minutes after lens settling of study lens.(Upgaze Lag and Post-blink Movement in mm)
Time Frame: Day 2 - 30 minutes
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: lens
Arm/Group | F55 SPHERE LENS P1 | F55 ASPHERE LENS P1 | F55 SPHERE LENS P2 | BF SPHERE LENS P2 | PCM SPHERE LENS P3 | BF SPHERE LENS P3
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Number analyzed (lens) | 20 | 20 | 20 | 20 | 20 | 20
millimeters
  Upper Gaze Lag | 0.11 (0.45) | 0.14 (0.45) | 0.13 (0.38) | 0.05 (0.16) | 0.33 (0.73) | 0.00 (0.00)
  Post-blink Movement | 0.32 (0.25) | 0.33 (0.22) | 0.31 (0.35) | 0.23 (0.21) | 0.39 (0.42) | 0.25 (0.20)

28. Primary Outcome: Investigator Fit Preference Contact Lens 30 Minutes Wear (Day 1 Study Lenses - Pair 1)
Description: Investigator rating of fit preference upon contact lens settling of pair 1. Collected at 30 minutes post settling for each lens. Percent of investigators that strongly prefer lens or have No Preference. (forced choice preference for right or left eye; Strong R, Slight R, No Pref, Slight L, Strong L)
Time Frame: Day 1- 30 minutes
Measure: Number; unit: percentage of investigators
Units Other Than Participants: eyes
Arm/Group | B55 SPHERE LENS P1 / B55 PREMIER ASPHERE LENS P1
Number analyzed (Participants) | 20
Number analyzed (eyes) | 40
percentage of investigators
  B55 SPHERE LENS P1 | 5
  B55 PREMIER ASPHERE LENS P1 | 10
  No Preference | 85

29. Primary Outcome: Investigator Fit Preference Contact Lens 30 Minutes Wear (Day 1 Study Lenses - Pair 2)
Description: Investigator rating of fit preference upon contact lens settling of pair 2. Collected at 30 minutes post settling for each lens. Percent of investigators that strongly prefer lens or have No Preference. (forced choice preference for right or left eye; Strong R, Slight R, No Pref, Slight L, Strong L)
Time Frame: Day 1- 30 minutes
Measure: Number; unit: percentage of investigators
Units Other Than Participants: eyes
Arm/Group | B55 SPHERE LENS P2 / AV SPHERE LENS P2
Number analyzed (Participants) | 20
Number analyzed (eyes) | 40
percentage of investigators
  B55 SPHERE LENS P2 | 15
  AV SPHERE LENS P2 | 5
  No Preference | 80

30. Primary Outcome: Investigator Fit Preference Contact Lens 30 Minutes Wear (Day 1 Study Lenses - Pair 3)
Description: Investigator rating of fit preference upon contact lens settling of pair 3. Collected at 30 minutes post settling for each lens. Percent of investigators that strongly prefer lens or have No Preference. (forced choice preference for right or left eye; Strong R, Slight R, No Pref, Slight L, Strong L)
Time Frame: Day 1 - 30 minutes
Measure: Number; unit: percentage of investigators
Units Other Than Participants: eyes
Arm/Group | B55 SPHERE LENS P3 / BF SPHERE LENS P3
Number analyzed (Participants) | 20
Number analyzed (eyes) | 40
percentage of investigators
  B55 SPHERE LENS P3 | 5
  BF SPHERE LENS P3 | 10
  No Preference | 85

31. Primary Outcome: Investigator Fit Preference Contact Lens 30 Minutes Wear (Day 2 Study Lenses - Pair 1)
Description: as for outcome 28
Time Frame: Day 2 - Insertion
Measure: Number; unit: percentage of investigators
Arm/Group | F55 SPHERE LENS P1 / F55 PREMIER ASPHERE LENS P1
Number analyzed (Participants) | 20
percentage of investigators
  F55 SPHERE LENS P1 | 5
  F55 PREMIER ASPHERE LENS P1 | 5
  No Preference | 90

32. Primary Outcome: Investigator Fit Preference Contact Lens 30 Minutes Wear (Day 2 Study Lenses - Pair 2)
Description: as for outcome 29
Time Frame: Day 2 - Insertion
Measure: Number; unit: percentage of investigators
Arm/Group | F55 SPHERE LENS P2 / BIOFINITY LENS P2
Number analyzed (Participants) | 20
percentage of investigators
  F55 SPHERE LENS P2 | 10
  BIOFINITY LENS P2 | 40
  No Preference | 50

33. Primary Outcome: Investigator Preference Contact Lens 30 Minutes Wear (Day 2 Study Lenses - Pair 3)
Description: as for outcome 30
Time Frame: Day 2 - Insertion
Measure: Number; unit: percentage of investigators
Arm/Group | PCM SPHERE LENS P3 / BF SPHERE LENS P3
Number analyzed (Participants) | 20
percentage of investigators
  PCM SPHERE LENS P3 | 5
  BF SPHERE LENS P3 | 35
  No Preference | 60

34. Primary Outcome: Overall Ease of Lens Handling (Day 1 Study Lenses)
Description: Participant rating of overall lens handling regarding insertion and removal. Collected at post-removal for each lens on Day 1. (0-100, 0=very difficult, 100=very easy
Time Frame: Day 1 - After Removal
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | B55 SPHERE LENS P1 | B55 PREMIER ASPHERE LENS P1 | B55 SPHERE LENS P2 | AV SPHERE LENS P2 | B55 SPHERE LENS P3 | BF SPHERE LENS P3
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
units on a scale | 95 (10) | 95 (10) | 95 (10) | 93 (12) | 94 (9.3) | 92 (15.4)

35. Primary Outcome: Overall Ease of Lens Handling (Day 2 Study Lenses)
Description: Participant rating of overall lens handling regarding insertion and removal. Collected at post-removal for each lens on Day 2. (0-100, 0=very difficult, 100=very easy
Time Frame: Day 2 - After Removal
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | F55 SPHERE LENS P1 | F55 ASPHERE LENS P1 | F55 SPHERE LENS P2 | BF SPHERE LENS P2 | PCM SPHERE LENS P3 | BF SPHERE LENS P3
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
units on a scale | 96 (7.6) | 96 (8.1) | 96 (9.8) | 94 (12) | 94 (16) | 94 (16)

ADVERSE EVENTS:
Time Frame: From dispense up to day 2 for both lenses
Arm/Group | Pair 1 (Ocufilcon D / Ocufilcon D) | Pair 2 (Ocufilcon D / Enfilcon A) | Pair 3 (Ocufilcon D / Comfilcon A) | Pair 4 (Methafilcon A / Methafilcon A) | Pair 5 (Methafilcon A / Comfilcon A) | Pair 6 (Omafilcon A / Comfilcon A)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior consent from the sponsor.